CLINICAL TRIAL: NCT02402946
Title: Valoración Objetiva y Tratamiento de la rumiación
Brief Title: Placebo-controlled, Randomized Trial of a Simplified Biofeedback Technique for the Treatment of Rumination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)200/2011 ammendment
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2016-11

CONDITIONS: Rumination Disorders
MeSH Terms: conditions — Rumination Syndrome | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback (Experimental): Abdomino-thoracic muscle activity after a challenge meal will be recorded by EMG and the signal will be displayed on a monitor but not showed to the patients; in the biofeedback group, patients will be instructed to control, abdomino-thoracic muscle activity
  Interventions: Behavioral: Biofeedback
- Placebo medication (Placebo Comparator): Electromyography will be recorded but not shown to the patients. Patienst will take a pill of placebo and receive no instructions about controlling muscular activity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Biofeedback
  Arms: Biofeedback
Drug: Placebo
  Arms: Placebo medication

SUMMARY:
Rumination syndrome is characterized by effortless recurrent regurgitation of recently ingested food into the mouth, with consequent expulsión or re-chewing and swallowing. In a previous study we showed that rumination is produced by an unperceived, somatic response to food ingestión. After having identified the key mechanisms of rumination, we developed an original EMG guided biofeedback technique with specific targets for correction, based on EMG-guided control of abdomino-thoracic muscular activity, and in a pilot study we showed the potential effectivity of this treatment. In a subsequent study this technique was validated by a formal placebo-controlled, randomized trial. The current aim is to test the efficacy of a simplified biofeedback technique not requiring EMG-guided control.

DETAILED DESCRIPTION:
Abdomino-thoracic muscle activity after a challenge meal will be recorded by EMG: in the biofeedback group, patients will be instructed to control muscle activity, whereas in the placebo group patients will not. In each patient 3 sessions will be performed over a 10-day period. Physiological (muscular activity by EMG) and clinical outcomes (number of rumination events by questionnaries administered daily for 10 days) will be measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Rumination syndrome

Exclusion Criteria:

* relevant organic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of regurgitation episodes | 28 days

SECONDARY OUTCOMES:
Postprandial abdominal symptoms | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — Hospital Universitary vall d'Hebron
Locations (2):
- Spain (2):
  - University Hospital Vall d'Hebron, Barcelona, Catalonia
  - Fernando Azpiroz, Barcelona

REFERENCES:
- [Background] Barba E, Burri E, Accarino A, Malagelada C, Rodriguez-Urrutia A, Soldevilla A, Malagelada JR, Azpiroz F. Biofeedback-guided control of abdominothoracic muscular activity reduces regurgitation episodes in patients with rumination. Clin Gastroenterol Hepatol. 2015 Jan;13(1):100-6.e1. doi: 10.1016/j.cgh.2014.04.018. Epub 2014 Apr 24. PMID 24768808